CLINICAL TRIAL: NCT03421145
Title: A Prospective, Randomized, Blinded, Clinical Study to Evaluate Effects of an Oral Rinse on Plaque and Gingivitis
Brief Title: A Clinical Study to Evaluate Effects of an Oral Rinse on Plaque and Gingivitis
Status: Completed | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EM-11-050003
Record Dates: First submitted 2017-12-20; First posted 2018-02-05 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Plaque
Keywords: Dental Plaque
MeSH Terms: conditions — Plaque, Amyloid; Dental Plaque | interventions — Water

STUDY DESIGN:
Intervention Model Description: prospective, randomized, blinded, clinical study to evaluate an oral rinse on plaque and gingivitis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Principal Investigator and clinical examiners will be blinded to the treatment products. No clinical examiners will see the allocated rinse assigned per the randomization schedule.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (4):
- 3M™ Oral Rinse (Experimental): Subjects assigned to the Experimental Oral Rinse ('Plaque control device) will swish a volume of 15 mL of the Experimental Rinse for 30 seconds followed by expectoration, twice a day (morning and evening), after brushing teeth, for the 6-month duration of the study. They will use the dosing cup provided by the study team to ensure that the proper dose of rinse is used. Subjects will be instructed not to eat or drink for 30 minutes after using the rinse and to complete the subject daily diary.
  Interventions: Device: 3M™ Oral Rinse
- Vehicle Control Oral Rinse (Placebo Comparator): Vehicle control oral rinse (no active ingredient). Subjects assigned to the Placebo Comparator will swish a volume of 15 mL of the Placebo Comparator rinse for 30 seconds followed by expectoration, twice a day (morning and evening), after brushing teeth, for the 6-month duration of the study. They will use the dosing cup provided by the study team to ensure that the proper dose of rinse is used. Subjects will be instructed not to eat or drink for 30 minutes after using the rinse and to complete the subject daily diary.
  Interventions: Other: Vehicle Control Oral Rinse
- PerioShield™ Oral Health Rinse (Active Comparator): Active control predicate device oral rinse ('Plaque control agent') Subjects assigned to the Active Comparator will swish a volume of 10 mL of the Active Comparator rinse for 30 seconds followed by expectoration, twice a day (morning and evening), after brushing teeth, for the 6-month duration of the study. They will use the dosing cup provided by the study team to ensure that the proper dose of rinse is used. Subjects will be instructed not to eat or drink for 30 minutes after using the rinse and to complete the subject daily diary.
  Interventions: Device: PerioShield™ Oral Health Rinse
- Water (Sham Comparator): Water sham control oral rinse (not a Plaque control agent) Subjects assigned to the Sham Comparator will swish a volume of 15 mL of the Sham Comparator rinse for 30 seconds followed by expectoration, twice a day (morning and evening), after brushing teeth, for the 6-month duration of the study. They will use the dosing cup provided by the study team to ensure that the proper dose of rinse is used. Subjects will be instructed not to eat or drink for 30 minutes after using the rinse and to complete the subject daily diary.
  Interventions: Other: Water

INTERVENTIONS:
Device: 3M™ Oral Rinse — The Investigational Rinse contains a sugar-based surfactant using a proprietary formula. The intended use of the product is to help prevent and reduce plaque accumulation on the teeth and related gum-tissue inflammation (gingivitis).
  Other Names: Plaque control device
  Arms: 3M™ Oral Rinse
Other: Vehicle Control Oral Rinse — The Placebo Comparator oral rinse is similar to the Experimental Oral Rinse only it does not contain the active ingredient.
  Other Names: Placebo Comparator
  Arms: Vehicle Control Oral Rinse
Device: PerioShield™ Oral Health Rinse — PerioShield™ Oral Health Rinse (0.2% delmopinol hydrochloride) is marketed in the US and was purchased for use in this study.
  Other Names: Active Comparator
  Arms: PerioShield™ Oral Health Rinse
Other: Water — Purified bottled water containing no active ingredients.
  Other Names: Sham Comparator
  Arms: Water

SUMMARY:
Rinse contains an anti-plaque agent that helps prevent the accumulation of dental plaque associated with gingivitis.

DETAILED DESCRIPTION:
This is a prospective, single site, randomized, parallel, blinded clinical trial. Subjects will be randomly assigned to one of four treatment groups identified as Product A, Product B, Product C or Product D.

Subjects will be screened for eligibility and entered into a washout period that is at least 7 days, during which time they will be provided with study toothbrush, toothpaste and dental floss. No oral rinses or medication that alters oral tissue health will be used or taken during the washout period. After randomization, the designated rinse will be placed into a non-transparent container so that other subjects and clinical examiners do not see the allocated rinse per the randomization schedule.

Examinations for the clinical endpoints (PI, GI and BI) will be conducted at the baseline, 3-month, and 6-month visits.

Interim visits will be scheduled to review diary, replenish study supplies, check study compliance, etc. Subjects will be provided Colgate Regular toothpaste, dental floss and a soft toothbrush (replaced at 3 months) for use during the 6-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to whom these criteria apply will be entered into the 7-day washout

  * Able to understand and willing to sign the Informed Consent
  * In good general health ages 18 and older
  * Have at least 20 natural teeth, including at least one molar and one premolar in each quadrant but excluding the third molars
  * Willing to return to the study facility for scheduled study visits and recalls
  * Agree not to use other oral hygiene products (non-study toothpaste, dental floss, mouth rinse, chewing gum)
  * Agree not to brush or floss teeth after 10:00 pm the night before and not eat or drink 4 hours before an appointment
  * Agree to the study instructions and visit schedule, including no eating or drinking for 4 hours before assessment appointments

Subjects must meet the screening inclusion criteria and these additional requirements for enrollment:

* Completed the washout period (at least 7 days) using only the study toothbrush, dental floss and toothpaste
* A qualifying baseline GI of at least 1.0, as determined by the Löe-Silness Gingival Index (GI)
* A qualifying baseline Modified Quigley-Hein (Lobene-Soparkar Modification of Turesky's modification) Plaque Index (PI) of at least 1.5 Subjects will be excluded if they do not meet the screening exclusion criteria.

Exclusion Criteria:

* Subjects to whom these conditions apply will be excluded:

  * A history of antibiotic therapy within the previous 30 days or have a condition that is likely to need antibiotic treatment over the course of the study (eg, cardiac conditions requiring antibiotic prophylaxis such as heart murmurs, pacemakers, or prosthetic heart valves, and prosthetic implants)
  * A history of using antimicrobial oral mouth rinse during the past 3 months
  * Taking medications which may alter gingival appearance/bleeding
  * Use of anticonvulsants, calcium channel blockers, or other medications with side effects known to impact oral health
  * Current participation in any other clinical study within the past 30 days
  * Reside in the same household with a subject already enrolled in the study
  * Dry mouth due to head/neck radiation therapy
  * Orthodontic appliances
  * Widespread caries or chronic neglect
  * Gross pathological changes of oral soft tissues
  * Known history of sensitivity to oral hygiene products
  * Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive alveolar bone loss)
  * Pregnant or nursing or plan to become pregnant within the 6 month study duration
  * Medical and oral conditions that, in the investigator's judgment, may compromise the subject's safety or interfere with the conduct and outcome of the study
  * Difficult to be compliant with study visits, such as extensive travel commitments or lack of transportation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda Dental Reserach, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parameter on plaque-induced gingivitis. American Academy of Periodontology. J Periodontol. 2000 May;71(5 Suppl):851-2. doi: 10.1902/jop.2000.71.5-S.851. PMID 10875689
- [Background] 2. National Institute of Health and Clinical Excellence (NICE). Dental recall interval between routine dental examinations. http://guidance.nice.org.uk/CG19 Clinical Guideline 19; 2004.
- [Background] Baehni PC, Takeuchi Y. Anti-plaque agents in the prevention of biofilm-associated oral diseases. Oral Dis. 2003;9 Suppl 1:23-9. doi: 10.1034/j.1601-0825.9.s1.5.x. PMID 12974527
- [Background] Moran JM. Chemical plaque control--prevention for the masses. Periodontol 2000. 1997 Oct;15:109-17. doi: 10.1111/j.1600-0757.1997.tb00110.x. No abstract available. PMID 9643238
- [Background] Steinberg D, Feldman M, Ofek I, Weiss EI. Effect of a high-molecular-weight component of cranberry on constituents of dental biofilm. J Antimicrob Chemother. 2004 Jul;54(1):86-9. doi: 10.1093/jac/dkh254. Epub 2004 May 26. PMID 15163648
- [Background] Li Y, Lee S, Hujoel P, Su M, Zhang W, Kim J, Zhang YP, DeVizio W. Prevalence and severity of gingivitis in American adults. Am J Dent. 2010 Feb;23(1):9-13. PMID 20437720
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Talbott K, Mandel ID, Chilton NW. Reduction of baseline gingivitis scores with repeated prophylaxes. J Prev Dent. 1977 Nov-Dec;4(6):28-9. No abstract available. PMID 275491
- [Background] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Lobene RR, Soparkar PM, Newman MB. Use of dental floss. Effect on plaque and gingivitis. Clin Prev Dent. 1982 Jan-Feb;4(1):5-8. No abstract available. PMID 6980082
- [Background] Caton JG, Polson AM. The interdental bleeding index: a simplified procedure for monitoring gingival health. Compend Contin Educ Dent (Lawrenceville). 1985 Feb;6(2):88, 90-2. No abstract available. PMID 3871687
- [Background] 13. FDA FOI, 510(k) for Sinclair Pharmaceuticals PMA for Decapinol, Retrieved from http://www.fda.gov/downloads/AboutFDA/CentersOffices/CDRH/CDRHFOIAElectronicReadingRoom/UCM237296.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects entered a washout phase after meeting screening qualifications. These subjects used the study oral hygiene supplies (toothpaste, toothbrush, and dental floss) for at least 7 days before the baseline qualification visit. Subjects were randomized to enter the study after their baseline qualifications were met.
Period: Overall Study
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Started | 50 | 50 | 50 | 50
Completed | 47 | 48 | 45 | 47
Not Completed | 3 | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 49 | 47 | 46 | 189
  >=65 years | 3 | 1 | 3 | 4 | 11
Age, Continuous [Median (Full Range); unit: years] | 37 [18 to 67] | 37 [23 to 67] | 37 [20 to 76] | 38 [19 to 72] | 37 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 21 | 21 | 80
  Male | 31 | 31 | 29 | 29 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 17 | 19 | 69
  Not Hispanic or Latino | 35 | 32 | 33 | 31 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 8 | 9 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 11 | 6 | 5 | 5 | 27
  White | 32 | 33 | 35 | 34 | 134
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 2 | 0 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 50 | 50 | 200
Plaque Index Score [Mean (Standard Deviation); unit: score on a scale] | 2.725 (0.4953) | 2.641 (0.47) | 2.702 (0.4986) | 2.82 (0.5597) | 2.722 (0.5073)
Gingivitis Index Score [Mean (Standard Deviation); unit: score on a scale] | 1.277 (0.1793) | 1.247 (0.1521) | 1.237 (0.13) | 1.277 (0.2016) | 1.259 (0.1676)
Bleeding Index Score [Mean (Standard Deviation); unit: score on a scale] | 0.452 (0.2388) | 0.413 (0.2203) | 0.399 (0.196) | 0.426 (0.2459) | 0.422 (0.2253)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index Score Per Participant at 6 Months
Description: Modified Quigley-Hein Plaque Index 0 = No plaque
  1. = Separate flecks of plaque at the cervical margin of the tooth
  2. = A thin, continuous band of plaque (up to one mm) at the cervical margin of the tooth.
  3. = A band of plaque wider than 1 mm, but covering less than 1/3 of the crown of the tooth.
  4. = Plaque covering at least 1/3, but less than 2/3 of the crown of the tooth.
  5. = Plaque covering 2/3 or more of the crown of the tooth. Each tooth is scored for supragingival plaque on six surfaces: 1) mesio-facial; 2) mid-facial; 3) disto-facial; 4) mesio-lingual; 5) mid-lingual; and 6) disto-lingual. Third molars and those teeth with cervical restorations or prosthetic crowns will be excluded from the scoring procedure.
  The PI score of the individual can be obtained by adding the scores of all surfaces and dividing by the number of surfaces examined.
Time Frame: 6 months
Population: study subjects who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 47 | 48 | 45 | 47
score on a scale | 2.12 (0.516) | 2.70 (0.453) | 2.23 (0.473) | 2.84 (0.469)
Statistical Analysis 1: Comparison: 3M™ Oral Rinse vs Vehicle Control Oral Rinse; Test type: Superiority; p < 0.0001, ANCOVA

2. Primary Outcome: Gingivitis Index Score Per Participant at 6 Months
Description: Löe-Silness Gingival Index
  0 = Absence of inflammation.
  1. = Mild inflammation: slight change in color and little change in texture.
  2. = Moderate inflammation: moderate glazing, redness, edema, hypertrophy. Tendency to bleed upon probing.
  3. = Severe inflammation: marked redness and hypertrophy. Tendency to spontaneous bleeding.
  The gingival surface surrounding each tooth (all natural teeth) will be scored on six surfaces: 1) mesio-facial; 2) mid-facial; 3) disto-facial; 4) mesio-lingual; 5) mid-lingual; and 6) disto-lingual. Third molars and those teeth with cervical restorations or prosthetic crowns will be excluded from the scoring procedure. The GI score of the individual can be obtained by adding the scores of all surfaces and dividing by the number of surfaces examined.
Time Frame: 6 months
Population: Study subjects who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 47 | 48 | 45 | 47
score on a scale | 1.09 (0.173) | 1.29 (0.144) | 1.11 (0.155) | 1.32 (0.158)
Statistical Analysis 1: Comparison: 3M™ Oral Rinse vs Vehicle Control Oral Rinse; Test type: Superiority; p < 0.0001, ANCOVA

3. Secondary Outcome: Plaque Index Score Per Participant at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: Study subjects that presented for 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 48 | 48 | 46 | 48
score on a scale | 2.43 (0.501) | 2.79 (0.439) | 2.49 (0.613) | 2.85 (0.476)
Statistical Analysis 1: Comparison: 3M™ Oral Rinse vs Vehicle Control Oral Rinse; Test type: Superiority; p < 0.0001, ANCOVA

4. Secondary Outcome: Bleeding Assessment Per Participant at 6 Months
Description: Eastman Interdental Bleeding Index 0 = Absence of bleeding.
  1 = Presence of bleeding The interdental cleaner is inserted between two teeth from the facial aspect, depressing the interdental tissues 1 to 2 mm. This is repeated four times and the presence or absence of bleeding within 15 seconds is recorded. The absence or presence of bleeding will be recorded for each examined site (between two teeth), and a score will be calculated as the number of bleeding sites out of the number of examined sites for each evaluation on a subject.
Time Frame: 6 months
Population: Study subjects who presented for 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 47 | 48 | 45 | 47
score on a scale | 0.28 (0.198) | 0.42 (0.197) | 0.28 (0.174) | 0.43 (0.246)
Statistical Analysis 1: Comparison: 3M™ Oral Rinse vs Vehicle Control Oral Rinse; Test type: Superiority; p < 0.0001, ANCOVA

5. Secondary Outcome: Gingivitis Index Per Participant at 3 Months
Description: as for outcome 2
Time Frame: 3 months
Population: Study subjects who presented for 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 48 | 48 | 46 | 48
score on a scale | 1.17 (0.191) | 1.27 (0.163) | 1.19 (0.155) | 1.30 (0.164)
Statistical Analysis 1: Comparison: 3M™ Oral Rinse vs Vehicle Control Oral Rinse; Test type: Superiority; p < 0.0001, ANCOVA

6. Secondary Outcome: Bleeding Index Per Participant at 3 Months
Description: as for outcome 4
Time Frame: 3 months
Population: study subjects who presented for 3-month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
Number analyzed (Participants) | 48 | 48 | 46 | 48
score on a scale | 0.34 (0.229) | 0.40 (0.200) | 0.33 (0.139) | 0.40 (0.247)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 3M™ Oral Rinse | Vehicle Control Oral Rinse | PerioShield™ Oral Health Rinse | Water
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 32/50 | 16/50 | 43/50 | 10/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M™ Oral Rinse (N=50) | Vehicle Control Oral Rinse (N=50) | PerioShield™ Oral Health Rinse (N=50) | Water (N=50)
Dry Mouth (Gastrointestinal disorders) | 9 (9) | 10 (10) | 19 (19) | 3 (3)
Dry Throat (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 6 (6) | 3 (3) | 22 (22) | 2 (2)
Oral discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 7 (7) | 1 (1)
Oral hypo-aesthesia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 38 (38) | 1 (1) — numbness
Oral mucosal exfoliation (Gastrointestinal disorders) | 25 (25) | 1 (1) | 10 (10) | 0 (0) — tissue sloughing
Tooth sensitivity (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 1 (1) — inflammation
Chapped Lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oral paraesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — tingling of mouth
Root canal infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — drooling
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol with planned Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT03421145/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT03421145/SAP_001.pdf